CLINICAL TRIAL: NCT04894617
Title: Amantadine for COVID-19: A Randomized, Placebo Controlled, Double-blinded, Clinical Trial
Brief Title: Amantadine for COVID-19
Acronym: ACT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Nina Weis, Professor, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02032021; 2021-001177-22 (EudraCT Number)
Record Dates: First submitted 2021-05-12; First posted 2021-05-20 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Amantadine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Unblinded personnel will perform randomization into one of two arms (ratio 1:1). The randomization list will be generated centrally in random blocks. Blinded personnel will not have access to the randomization key. Unblinded staff will deliver sealed envelopes containing treatment allocation to blinded study personnel to use for emergency unblinding.
  All investigators, outcome assessors, and study participants will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amantadine (Active Comparator): The intervention group will receive a dose at day 1 of amantadine 100 mg followed by 100 mg amantadine after 6 hours. The following 4 consecutive days, study participants will receive a daily dose of 200mg amantadine, 100 mg (1 capsule) morning and 100 mg (1 capsule) evening, yielding 5 days of treatment in total (10 capsules in total).
  Interventions: Drug: Amantadine
- Placebo (Placebo Comparator): The control group will receive placebo treatment with lactose monohydrate; 1 capsule, followed by 1 capsule after 6 hours on day 1. The following 4 consecutive days, study participants will receive 1 capsule morning and 1 capsule evening, yielding 5 days of treatment in total (10 capsules in total).
  Interventions: Drug: Lactose monohydrate

INTERVENTIONS:
Drug: Amantadine — 200 mg Amantadine daily for a total of 5 days.
  Arms: Amantadine
Drug: Lactose monohydrate — Lactose monohydrate two tablet daily for a total of 5 days.
  Arms: Placebo

SUMMARY:
Introduction:

Corona virus disease 19 (COVID-19) is a devastating pandemic. By early February 2021, more than 102 million people were infected globally with more than 2.2 million reported deaths. Current treatments are approved for hospitalized patients with severe COVID-19 only. No treatment is approved to prevent progression to severe COVID-19 in the early stages of disease. Previous studies have indicated that amantadine is effective against severe acute respiratory syndrome corona virus 1 (SARS-CoV-1). Trials are needed to determine if this translates to a beneficial effect in patients with COVID-19. We hypothesize that preemptive therapy with amantadine of non-hospitalized high-risk adults with SARS-CoV-2 infection disease will prevent disease progression and hospitalization.

Methods and analysis:

The study is a randomized, double-blinded, placebo-controlled, single center study with two treatment arms; oral amantadine or placebo. Individuals with confirmed SARS-CoV-2 infection and one of following; i) age ≥ 40 years or ii) ≥ 18 years of age with at least one comorbidity or iii) ≥ 18 years of age with a body mass index (BMI) above 30 will be enrolled in the study. We plan to enroll 121 persons in each arm, with a total of 242 participants. Follow up period is 90 days. The primary outcome is disease severity on day 14 assessed by the 8-point COVID outcome scale proposed by the world health organization.

Ethics and dissemination:

Approvals by the Ethics Committee and National Competent Authorities will be obtained prior to study initiation. Results will be submitted for publication in a peer-reviewed journal and presented at international conferences.

Impact:

The results of the study will contribute with important knowledge on the efficacy and safety of oral amantadine in the treatment of non-hospitalized high-risk individuals with SARS-CoV-2 infection.

DETAILED DESCRIPTION:
BACKGROUND

Globally, Corona virus disease 19 (COVID-19) has caused more than 2.2 million deaths.

Most infected cases present with mild respiratory symptoms and fever, and spontaneously recover within two weeks. However, for approximately 20% of the cases, the disease will progress to pneumonia and in the most severe cases respiratory failure, multiple organ dysfunction, and death. Individuals aged ≥ 50 years of age and adults with known comorbidity or obesity are at particular risk of a severe course of the disease.

Within the past year treatments have proven to be beneficial for severe COVID-19 in randomized controlled trials. However, no treatment has been proven to inhibit progression from mild to severe COVID-19. Such a treatment could potentially have major impact on long-term morbidity and mortality especially in areas with limited access to vaccines. The fastest way of identifying such a treatment may be repurposed drugs. Other benefits of repurposed drugs include affordable prices and known safety profiles.

Amantadine is a potential treatment candidate that for years has been employed in the clinic for treatment of influenza virus A infection and for treatment of dyskinesia associated with Parkinson's disease. Furthermore, a potential repurposing of amantadine for the prevention and treatment of severe acute respiratory syndrome corona virus(SARS CoV-2) infection has been suggested. Two viroporins have been identified in the genome of SARS-CoV-2, Protein E and Protein 3a, with strong similarities to the viroporins in the deadly coronavirus SARS-CoV-1. The expression of both Protein E and 3a has been shown to promote SARS-CoV-1 replication and virulence, and the deletion of SARS CoV-1 protein E gene attenuates the virus. Amantadine has previously been shown to bind and inhibit protein E. Knocking down E protein ion channel activity in SARS CoV-1 decreases edema accumulation, which is the major determinant of acute respiratory distress syndrome (ARDS). Furthermore, levels of inflammasome-activated interleukin-1b, tumor necrosis factor (TNF) and interleukin-6 were reduced in the lung airways of the animals infected with viruses lacking E protein ion channel activity, indicating that E protein ion channel function is required for inflammasome activation. All these key cytokines promote the progression of lung damage and ARDS pathology. As such, by potentially blocking protein E ion channel activity, amantadine may prevent severe progression of SARS-CoV-2. Thus, we hypothesize that amantadine can ameliorate disease progression in persons with SARS-CoV-2 infection.

OBJECTIVES The aim of the study is to investigate if early preemptive therapy with amantadine in non-hospitalized high-risk adult individuals with COVID-19 disease can limit disease progression.

DESIGN This is a randomized, double-blinded, placebo-controlled study comparing amantadine with placebo 1:1. Follow up is 90 days in total, with close follow up during the first 14 days, and severe adverse events (SAE) monitoring throughout the study period.

Persons who test positive for SARS-CoV-2 by polymerase chain reaction (PCR)-testing will be identified through lists from laboratories performing the tests and recruited through invitation letters as well as online advertisement. If they fulfill all of the inclusion criteria and none of the exclusion criteria and choose to consent to enrollment after thorough oral and written information, they will proceed to randomization.

RANDOMIZATION AND BLINDING Unblinded personnel at the regional pharmacy will perform randomization into one of two arms (ratio 1:1). The randomization list will be generated centrally in random blocks. Blinded personnel will not have access to the randomization key. All investigators, outcome assessors, and study participants will be blinded to the treatment allocation.

Emergency unblinding can be performed if necessary, for the welfare of the study participant. Efforts should be made to avoid unblinding. If the treatment of a patient has been unblinded, the treatment course must be discontinued, but the patient will still be subject to follow up.

DATA COLLECTION AND FOLLOW-UP Data collection will be a combination of assessments by a physician, trained medical student or nurse at day 1 and 7 and self-reporting, using online questionnaires at day 2-6, 14, 28 and 90. Study participants will be followed for a total of 90 days. Moreover, data will be retrieved from medical files and the Danish national patient registry and the civil registrations system.

WITHDRAWAL Apart from the participant's own withdrawal of written consent, participants will be withdrawn from the study if the investigator finds it necessary due to the participant safety. Safety reasons comprise any unintended serious adverse event related to the treatment.

No participants will be registered as lost to follow up. Protocol violation will be reported if participants do not receive the full dose of study drug, or fail to answer one or more of the questionnaires, unless the patient has been admitted to hospital.

TREATMENT

Both active treatments and placebo treatment will be prepared, packaged and labeled by pharmacists at the pharmacy of the Capital region in Denmark. To assure full blinding for both participants and investigators all treatment will be covered in non-transparent identical capsules.

Treatment adherence will be assessed through the daily web-based questionnaires on day 2-6 and by collection of the empty medicine box at assessment on day 7.

Amantadine Participants randomized to active treatment with amantadine will receive a daily dose of 200 mg amantadine with 100 mg (1 capsule) two times a day for a total of five days. Patients with reduced renal function (estimated glomerular filtration rate (eGFR 35-60 ml/min)) will receive the same dose on day one, but from day 2-5 a reduced dose of 100 mg once a day (daily dose 100mg) will be administered. Safety of amantadine is well tested for treatment and prophylaxis of influenza A at 200 mg a day for up to six weeks. Amantadine has a half-life of 17 hours.

Participants randomized to receive placebo will receive non-active lactose monohydrate oral placebo capsules. The number of placebo capsules are equal to the number of amantadine capsules.

EXPECTED RISKS AND BENEFITS Amantadine has previously been used in the treatment of Influenza A and has been shown to reduce Influenza A virus shedding and shorten the duration of symptoms by about a third, if administered early.

Current in vitro studies indicate that similar properties may be present against SARS-CoV-2. An older study has shown an effect of amantadine on coronaviruses and a recent study proposes that amantadine can be used to mitigate the effect of SARS-CoV-2.

As amantadine could potentially disrupt the lysosomal pathway, decrease the replication of SARS-CoV-2 as well as virus induced inflammation in SARS-CoV-2 positive patients, it may serve as a potent therapeutic leading to better clinical outcomes.

The most common side effects of amantadine include nausea, dizziness (lightheadedness), and insomnia. Blurry vision and/or impaired mental acuity may occur. Less frequently (1 to 5%) reported adverse reactions are: Depression, anxiety and irritability, hallucinations, confusion, anorexia, dry mouth, constipation, ataxia, livedo reticularis, peripheral edema, orthostatic hypotension, headache, somnolence, nervousness, dream abnormality, agitation, dry nose, diarrhea and fatigue.

DATA HANDLING Oral and written consent, including medical record access, must be given by the participant at the initial assessment. Once the informed consent is obtained, investigators, sponsor, representatives of the sponsor and the relevant regulatory authorities will have direct access to the patient's medical record. Information in the medical record will be accessed to the extent that it is necessary for the completion of the study, as well as control including self-monitoring, quality control and monitoring by regulatory authorities.

Baseline data on day 1, SARS-CoV-2 PCR results on day 7, primary and secondary outcomes; all-cause mortality, need of mechanical ventilation, hospitalization are retrieved from medical records.

All data on participants will be registered and kept in a single electronic case report form (eCRF) under one study patient identification number (ID).

Sponsor and investigators are obliged to handle all data on study participants confidentially in accordance with the General Data Protection Regulation [21] and the Data Protection Act. The primary investigator is responsible for completing eCRFs for all trial participants. At the end of the study, the primary investigator will extract data from the electronic database in order to perform the planned analyses on primary and secondary outcomes. Study data will subsequently be published only in pseudonymous form.

STATISTICS

Sample size The primary endpoint is clinical status on day 14 on an eight point ordinal scale. The assumed probabilities of being in a certain clinical state on day 14 are shown below. If we want to detect an odds ratio for a higher ordinal scale score of 0.5 with placebo as reference group and a simulated power of 80% a target sample size of 121 patients per arm is needed. Thus, a total sample size of 242 participants is required. Rates of hospitalization, oxygen requirement, mechanical ventilation, organ support and mortality are estimated based on epidemiological COVID-19 data reported from the Danish Serum Institute and descriptive studies from Denmark, California and Iceland.

Descriptor Score Probability No limitations to activities. 1 0.526 Limitations to activities. 2 0.354 Hospitalized no oxygen therapy. 3 0.028 Oxygen by mask or nasal prongs. 4 0.048 Non-invasive ventilation or high flow oxygen. 5 0.028 Intubation and mechanical ventilation. 6 0.012 Ventilation + additional organ support, 7 0.004 Extra corporal membrane oxygenation (ECMO) Death. 8 0.000

Statistical analysis of data Normally distributed continuous variables are presented as mean with standard deviation and t-tests are applied. Non-normally distributed continuous variables are presented as median with 25% and 75% quantiles and Mann-Whitney tests are applied.

Categorical data are presented as counts with frequencies. For categorical data we use chi-square test if cell counts are above 5 and Fisher's exact test or simulation if cells are below 5. The primary endpoint will be assessed using a proportional odds model adjusting for age, sex, Charlson's comorbidity index (CCI) and vaccination. The primary analysis will be intention to treat, however we will also provide a per protocol analysis.

All tests are done at a significance level of 0.05.

PUBLICATION

Positive, inconclusive as well as negative outcomes of the study will be published. The study will be registered at www.clinicaltrials.gov and www.clinicaltrialregister.eu prior to initiation. Additionally, trial results will be up-loaded to EudraCT as soon as possible, and no later than 1 year after trial completion. Data will subsequently be published at www.clinicaltrialregister.eu.

FUNDING The initiative for this study was taken by the sponsor, and medical doctors at the Departments of Infectious Diseases at Hvidovre Hospital. The study is a cooperation between researchers in the two institutions. The study will be set up and completed by staff at Departments of Infectious Diseases at Hvidovre Hospital. The sponsor has provided the idea for the study, background knowledge of the effects of amantadine on SARS-CoV-2 and has achieved funding from a private fund. The study is funded with 2.000.000 DKK from the private foundation BioInnovation Institute (BII). Study participants and the Research Ethics Committee of the Capital Region of Denmark will be informed, if additional funding has been granted.

Sponsor and investigators are independent of economic or competing interests. Participants will not be financially reimbursed. Results from the study are only for scientific and public use and have no commercial interest.

ELIGIBILITY:
Inclusion Criteria:

* Population at risk of developing severe COVID-19, defined as either:

  * Age ≥ 40 years
  * Age ≥ 18 years and at least one of the following comorbidities: Chronic heart disease without heart failure or proarrhythmic conditions or ventricular arrythmias, diabetes, chronic lung disease, hypertension, chronic kidney disease estimated glomerula filtration rate (GFR)<60 ml/minute, BMI

    * 30 kg/m2.
* COVID-19 disease confirmed by the presence of SARS-CoV-2 nucleic acid by polymerase chain reaction (PCR) within 5 days prior to inclusion.
* For women of childbearing age (defined as non-sterile premenopausal women):

Negative pregnancy test and willingness to use contraceptive during the study period (90 days)

● Provision of informed consent.

Exclusion Criteria:

* Current hospitalization
* Allergy to amantadine hydrochloride, rimantadine or inactive ingredients.
* Known history of:

  * Untreated narrow-angle glaucoma
  * Kidney disease with eGFR < 35 ml/min
  * Heart failure, proarrhythmic conditions, ventricular arrhythmias.
  * Seizures
  * Parkinson's disease
  * Gastric ulcer
  * Liver Disease
  * Hereditary galactose intolerance, lactose intolerance or glucose/galactose malabsorption
* Current use of:

  * Neuroleptics/antipsychotics/ levodopa
  * Anticholinergics
  * Thiazides
* Concurrent malignancy requiring chemotherapy
* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Clinical status on day 14 | 14 days
  Clinical status on day 14 according to 8 point ordinal scale for clinical improvement.
  No limitations to activities=1, Limitations to activities=2, Hospitalized no oxygen therapy=3, Oxygen by mask or nasal prongs=4, Non-invasive ventilation or high flow oxygen=5, Intubation and mechanical ventilation=6, Ventilation + additional organ support, ECMO=7, Death=8.

SECONDARY OUTCOMES:
Mortality | Day 7, 14, 28 and 90
  Mortality rate
Mechanical ventilation | Day 7, 14, 28 and 90
  Incidence of Mechanical ventilation
Hospitalization | Day 7, 14, 28 and 90
  Incidence of hospitalization
Duration of hospitalization | 90 days
  Duration of hospitalization
PCR SARS-CoV-2 | Day 7
  Proportion with negative SARS-CoV-2 oropharyngeal swap
Adverse events | 90 days
  Frequency of adverse events
Severe adverse events | 90 days
  Frequency of severe adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Nina M Weis, PhD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Background] DIMITROVA EK. Veklury. Eur Med Agency 2020. https://www.ema.europa.eu/en/medicines/human/EPAR/veklury (accessed February 3, 2021).
- [Background] Research C for DE and. FDA's approval of Veklury (remdesivir) for the treatment of COVID-19-The Science of Safety and Effectiveness. FDA 2020.
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Weekly epidemiological update - 2 February 2021 n.d. https://www.who.int/publications/m/item/weekly-epidemiological-update---2-february-2021 (accessed February 3, 2021)
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440
- [Background] WHO Rapid Evidence Appraisal for COVID-19 Therapies (REACT) Working Group; Sterne JAC, Murthy S, Diaz JV, Slutsky AS, Villar J, Angus DC, Annane D, Azevedo LCP, Berwanger O, Cavalcanti AB, Dequin PF, Du B, Emberson J, Fisher D, Giraudeau B, Gordon AC, Granholm A, Green C, Haynes R, Heming N, Higgins JPT, Horby P, Juni P, Landray MJ, Le Gouge A, Leclerc M, Lim WS, Machado FR, McArthur C, Meziani F, Moller MH, Perner A, Petersen MW, Savovic J, Tomazini B, Veiga VC, Webb S, Marshall JC. Association Between Administration of Systemic Corticosteroids and Mortality Among Critically Ill Patients With COVID-19: A Meta-analysis. JAMA. 2020 Oct 6;324(13):1330-1341. doi: 10.1001/jama.2020.17023. PMID 32876694
- [Background] Jefferson T, Demicheli V, Di Pietrantonj C, Rivetti D. Amantadine and rimantadine for influenza A in adults. Cochrane Database Syst Rev. 2006 Apr 19;2006(2):CD001169. doi: 10.1002/14651858.CD001169.pub3. PMID 16625539
- [Background] Smieszek SP, Przychodzen BP, Polymeropoulos MH. Amantadine disrupts lysosomal gene expression: A hypothesis for COVID19 treatment. Int J Antimicrob Agents. 2020 Jun;55(6):106004. doi: 10.1016/j.ijantimicag.2020.106004. Epub 2020 Apr 30. PMID 32361028
- [Background] DeDiego ML, Nieto-Torres JL, Regla-Nava JA, Jimenez-Guardeno JM, Fernandez-Delgado R, Fett C, Castano-Rodriguez C, Perlman S, Enjuanes L. Inhibition of NF-kappaB-mediated inflammation in severe acute respiratory syndrome coronavirus-infected mice increases survival. J Virol. 2014 Jan;88(2):913-24. doi: 10.1128/JVI.02576-13. Epub 2013 Nov 6. PMID 24198408
- [Background] Castano-Rodriguez C, Honrubia JM, Gutierrez-Alvarez J, DeDiego ML, Nieto-Torres JL, Jimenez-Guardeno JM, Regla-Nava JA, Fernandez-Delgado R, Verdia-Baguena C, Queralt-Martin M, Kochan G, Perlman S, Aguilella VM, Sola I, Enjuanes L. Role of Severe Acute Respiratory Syndrome Coronavirus Viroporins E, 3a, and 8a in Replication and Pathogenesis. mBio. 2018 May 22;9(3):e02325-17. doi: 10.1128/mBio.02325-17. PMID 29789363
- [Background] Current status of amantadine and rimantadine as anti-influenza-A agents: memorandum from a WHO meeting. Bull World Health Organ. 1985;63(1):51-6. PMID 3872736
- [Background] Nicholson KG, Wiselka MJ. Amantadine for influenza A. BMJ. 1991 Feb 23;302(6774):425-6. doi: 10.1136/bmj.302.6774.425. No abstract available. PMID 2004163
- [Background] Mathur A, Beare AS, Reed SE. In vitro antiviral activity and preliminary clinical trials of a new adamantane compound. Antimicrob Agents Chemother. 1973 Oct;4(4):421-6. doi: 10.1128/AAC.4.4.421. PMID 4364762
- [Background] Abreu GEA, Aguilar MEH, Covarrubias DH, Duran FR. Amantadine as a drug to mitigate the effects of COVID-19. Med Hypotheses. 2020 Jul;140:109755. doi: 10.1016/j.mehy.2020.109755. Epub 2020 Apr 25. PMID 32361100
- [Background] Haase N, Plovsing R, Christensen S, Poulsen LM, Brochner AC, Rasmussen BS, Helleberg M, Jensen JUS, Andersen LPK, Siegel H, Ibsen M, Jorgensen V, Winding R, Iversen S, Pedersen HP, Madsen J, Solling C, Garcia RS, Michelsen J, Mohr T, Mannering A, Espelund US, Bundgaard H, Kirkegaard L, Smitt M, Buck DL, Ribergaard NE, Pedersen HS, Christensen BV, Perner A. Characteristics, interventions, and longer term outcomes of COVID-19 ICU patients in Denmark-A nationwide, observational study. Acta Anaesthesiol Scand. 2021 Jan;65(1):68-75. doi: 10.1111/aas.13701. Epub 2020 Oct 3. PMID 32929715
- [Background] Lendorf ME, Boisen MK, Kristensen PL, Lokkegaard ECL, Krog SM, Brandi L, Brinth LS, Nolsoe RLM, Ryrso C, Eiken P, Bestle MH, Jorgensen IM, Pedersen-Bjergaard U, Lindegaard B, Christensen TB, Fischer TK. Characteristics and early outcomes of patients hospitalised for COVID-19 in North Zealand, Denmark. Dan Med J. 2020 Aug 12;67(9):A06200428. PMID 32800073
- [Background] Gudbjartsson DF, Helgason A, Jonsson H, Magnusson OT, Melsted P, Norddahl GL, Saemundsdottir J, Sigurdsson A, Sulem P, Agustsdottir AB, Eiriksdottir B, Fridriksdottir R, Gardarsdottir EE, Georgsson G, Gretarsdottir OS, Gudmundsson KR, Gunnarsdottir TR, Gylfason A, Holm H, Jensson BO, Jonasdottir A, Jonsson F, Josefsdottir KS, Kristjansson T, Magnusdottir DN, le Roux L, Sigmundsdottir G, Sveinbjornsson G, Sveinsdottir KE, Sveinsdottir M, Thorarensen EA, Thorbjornsson B, Love A, Masson G, Jonsdottir I, Moller AD, Gudnason T, Kristinsson KG, Thorsteinsdottir U, Stefansson K. Spread of SARS-CoV-2 in the Icelandic Population. N Engl J Med. 2020 Jun 11;382(24):2302-2315. doi: 10.1056/NEJMoa2006100. Epub 2020 Apr 14. PMID 32289214
- [Background] Myers LC, Parodi SM, Escobar GJ, Liu VX. Characteristics of Hospitalized Adults With COVID-19 in an Integrated Health Care System in California. JAMA. 2020 Jun 2;323(21):2195-2198. doi: 10.1001/jama.2020.7202. PMID 32329797
- [Background] The European Parliament and the Council of the European Union. General Data Protection Regulation. (2016) n.d.
- [Background] https://www.who.int/docs/default-source/coronaviruse/who-china-joint-mission-on-covid-19-final-report.pdf n.d
- [Background] Rodriguez-Morales AJ, Cardona-Ospina JA, Gutierrez-Ocampo E, Villamizar-Pena R, Holguin-Rivera Y, Escalera-Antezana JP, Alvarado-Arnez LE, Bonilla-Aldana DK, Franco-Paredes C, Henao-Martinez AF, Paniz-Mondolfi A, Lagos-Grisales GJ, Ramirez-Vallejo E, Suarez JA, Zambrano LI, Villamil-Gomez WE, Balbin-Ramon GJ, Rabaan AA, Harapan H, Dhama K, Nishiura H, Kataoka H, Ahmad T, Sah R; Latin American Network of Coronavirus Disease 2019-COVID-19 Research (LANCOVID-19). Electronic address: https://www.lancovid.org. Clinical, laboratory and imaging features of COVID-19: A systematic review and meta-analysis. Travel Med Infect Dis. 2020 Mar-Apr;34:101623. doi: 10.1016/j.tmaid.2020.101623. Epub 2020 Mar 13. PMID 32179124
- [Background] Sundhedsministeriet. Lov om klage- og erstatningsadgang inden for sundhedsvæsenet 2017